CLINICAL TRIAL: NCT04810611
Title: A Phase Ib, Multicenter, Open-label Platform Study of Select Drug Combinations in Adult Patients With Lower Risk (Very Low, Low, or Intermediate Risk) Myelodysplastic Syndrome
Brief Title: Phase Ib Study of Select Drug Combinations in Patients With Lower Risk MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453E12101; 2019-004623-21 (EudraCT Number)
Record Dates: First submitted 2021-03-09; First posted 2021-03-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic; myelodysplastic syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — sabatolimab; NIS-793; canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: MBG453 single agent (Experimental): Treatment with MBG453 single agent Q4W to confirm safety and tolerability of RD.
  Interventions: Drug: MBG453
- Arm 2: NIS793 single agent (Experimental): Treatment with NIS793 single agent Q3W to establish RD in this indication and confirm safety and tolerability.
  Interventions: Drug: NIS793
- Arm 3: canakinumab single agent (Experimental): Treatment with single agent canakinumab Q4W to confirm safety and tolerability of RD.
  Interventions: Drug: canakinumab
- Arm 4: MBG453 + NIS793 combination (Experimental): Treatment with combination of MBG453 and NIS793 Q3W to confirm safety and tolerability of combination RD.
  Interventions: Drug: MBG453; Drug: NIS793
- Arm 5: MBG453 + canakinumab combination (Experimental): Treatment with MBG453 + canakinumab combination Q4W to confirm safety and tolerability of combination RD.
  Interventions: Drug: MBG453; Drug: canakinumab

INTERVENTIONS:
Drug: MBG453 — Anti-TIM3 monoclonal antibody
  Other Names: sabatolimab
  Arms: Arm 1: MBG453 single agent; Arm 4: MBG453 + NIS793 combination; Arm 5: MBG453 + canakinumab combination
Drug: NIS793 — Anti-TGF-β monoclonal antibody
  Arms: Arm 2: NIS793 single agent; Arm 4: MBG453 + NIS793 combination
Drug: canakinumab — Anti-IL-1β monoclonal antibody
  Other Names: ACZ885
  Arms: Arm 3: canakinumab single agent; Arm 5: MBG453 + canakinumab combination

SUMMARY:
The purpose of this study was to characterize the safety, tolerability and confirm the dose for select single agents and combinations in patients with lower risk (very low, low, and intermediate risk) MDS.

DETAILED DESCRIPTION:
This was a phase Ib, multi center, open-label, platform study with multiple treatment arms.

The design of this study was adaptive to allow discontinuation of poorly tolerated or ineffective treatments and to facilitate the introduction of new candidate single agents or combinations. Study design included a dose escalation/confirmation part and a dose expansion.

The planned initial single agent and combination treatment arms were the following:

* Arm 1: MBG453 single agent
* Arm 2: NIS793 single agent
* Arm 3: canakinumab single agent
* Arm 4: MBG453 + NIS793 combination
* Arm 5: MBG453 + canakinumab combination Patients were treated in the dose confirmation/escalation part of the study in Arms 1, 2, 3 and 5. No patients were treated in Arm 4. The study did not progress into the expansion phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Patients must be ≥ 18 years of age at the time of signing the informed consent form (ICF).
3. Patients must have a diagnosis prior to participation in the study of IPSS-R very low, low, or intermediate risk MDS with ≤10% bone marrow blasts and one or more of the following:

   1. Symptomatic anemia with hemoglobin <10 g/dL that has relapsed after or is refractory to ESAs (or the patient is intolerant to ESAs)
   2. Symptomatic anemia with hemoglobin <10 g/dL) that is ESA-naive with EPO level ≥ 500 /uL
   3. Thrombocytopenia with platelets <30,000/uL or with clinically significant bleeding or bruising and platelets <50,000/uL
   4. Neutropenia with an absolute neutrophil count (ANC) <500/ µL or with recurrent and/or severe infections and an ANC that is <1000/ µL and amenable to response assessments by International Working Group (IWG) response criteria in myelodysplasia (Cheson et al 2006)
4. Patients who are refractory to, intolerant of, or ineligible/unable to receive SOC therapeutic options including lenalidomide
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
6. Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institutions' guidelines and be willing to undergo a bone marrow aspirate and/or biopsy at screening, during and at the end of therapy on this study -

Key Exclusion Criteria:

1. Systemic antineoplastic therapy (including cytotoxic chemotherapy, alpha-interferon, kinase inhibitors or other targeted small molecules, and toxin-immunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is longer, before the first dose of study treatment.
2. History of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes.
3. Patients with chronic myelomonocytic leukemia (CMML) or myelodysplastic/myeloproliferative neoplasms (MDS/MPN)
4. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF, M-CSF), thrombopoietin mimetics or ESAs anytime ≤ 2 weeks (or 5 half-lives, whichever is longer) prior to start of study treatment.
5. Systemic chronic corticosteroid therapy (>10 mg/day prednisone or equivalent) or any immunosuppressive therapy within 7 days of first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
6. For arms containing canakinumab: Patients with ANC < 500 /µL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Dose interruption reduction | 30 Months
  Dose tolerability
Incidence of DLTs | 30 Months
  Incidence of dose limiting toxicities (DLTs) during the first 2 cycle of treatment during the dose escalation/confirmation part
Dose intensity | 30 Months
  Dose tolerability
AE and SAE incidence | 30 months
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as per CTCAE v5.0, by treatment

SECONDARY OUTCOMES:
Reduction in red blood cell (RBC) / platelet transfusions from baseline in transfusion dependent patients | Baseline, 30 Months
  The number of red cell or platelet transfusions a patient receives over the course of study treatment will be compared to the patient's baseline transfusion requirements based on the number of transfusions received during the 16-weeks period prior to the start of study treatment.
Duration of transfusion independence lasting for >=8 weeks, >=12 weeks, >=16 weeks, >=24 weeks in transfusion dependent patients | 30 Months
  Red cell or platelet transfusion independence is defined as no red cell or platelet transfusions with a duration lasting for 8, 12, 16, or 24 weeks.
Change from baseline in hemoglobin (Hb) in transfusion dependent and transfusion independent patients | Baseline, 30 Months
  Hemoglobin levels over the course of the study will be compared to the patient's baseline level to monitor for improvements in anemia.
Change from baseline in platelet count in transfusion dependent and transfusion independent patients | Baseline, 30 Months
  Platelet count over the course of the study will be compared to the patient's baseline count to monitor for improvements in thrombocytopenia.
Change from baseline in Absolute Neutrophil Count/White Blood Cells (ANC/WBC) in transfusion dependent and transfusion independent patients | Baseline, 30 Months
  Platelet count over the course of the study will be compared to the patient's baseline count to monitor for improvements in thrombocytopenia.
Best Overall Response (BOR) in transfusion dependent and transfusion independent patients | 30 Months
  BOR is the best disease response recorded from the start of the treatment until disease progression/relapse. The subject's BOR will be calculated based on investigator's response evaluations per International Working Group (IWG) criteria.
Time to onset of transfusion independence in transfusion dependent patients | 30 Months
  Time to onset of either red cell transfusion independence or platelet transfusion independence.
Time to onset of BOR in transfusion dependent and transfusion independent patients | 30 Months
  Time to onset of BOR is defined as the time between date of start of study treatment to the date of first onset of Partial Response (PR) or better response.
Duration of Response (DOR) in transfusion dependent and transfusion independent patients | 30 Months
  DOR is defined as the duration from the first documented onset of complete response (CR), complete remission with partial hematologic recovery (CRh), bone marrow CR (mCR) or PR to the date of disease progression (PD) or relapse or death due to myelodysplastic syndrome (MDS).
Overall Response Rate (ORR) in transfusion dependent and transfusion independent patients | 30 Months
  ORR is the proportion of subjects with a best overall response of either CR or CRh, or mCR or PR.
Progression free survival (PFS) in transfusion dependent and transfusion independent patients | 30 Months
  PFS is defined as the time from the start of treatment until death due to any reason, disease progression, or relapse, whichever comes first.
Time to progression (TTP) in transfusion dependent and transfusion independent patients | 30 Months
  TTP is the time from the start of treatment to the date of PD, relapse or death due to underlying cancer.
Characterize pharmacokinetics for single agents and combinations: Cmax | 30 Months
  Serum concentrations and derived PK parameters
Characterize pharmacokinetics for single agents and combinations: Tmax | 30 Months
  Serum concentrations and derived PK parameters
Characterize pharmacokinetics for single agents and combinations: Ctrough | 30 Months
  Serum concentrations and derived PK parameters
Characterize the prevalence of immunogenicity | 30 Months
  Anti-drug antibody prevalence at baseline and on treatment.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - City Of Hope National Med Center Oncology, Duarte, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Massachusetts General Hospital ., Boston, Massachusetts
  - The Ohio State University Wexner Medical Center ., Columbus, Ohio
  - MD Anderson Cancer Center/University of Texas MD Anderson, Houston, Texas
- Novartis Investigative Site, Prahran, Victoria, Australia
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18275
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2574